CLINICAL TRIAL: NCT05996250
Title: Tolerance of an Immersive Virtual Reality Task Evaluating the Spatial Memory of Elderly Subjects and the Effects of Age, Gender and Level of Education on Performance
Brief Title: Tolerance of an Immersive Virtual Reality Task Evaluating the Spatial Memory of Elderly Subjects
Acronym: REVIAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL22_0203
Record Dates: First submitted 2023-08-01; First posted 2023-08-18 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Healthy Participants
Keywords: Virtual reality; ageing; spatial memory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immersive virtual reality task (Other): The immersive virtual reality task, specifically designed for this research, is an adaptation to humans of Morris Pool. The virtual environment is composed of a circular arena 22 virtual meters in diameter, delimited by a low wall. It features two visual landmarks and an invisible object to find. The activity includes a control training sequence, an evaluation sequence and a delayed recall performed approximately 20 minutes after the end of the evaluation sequence.
  The immersive reality task is performed once by the participants (the study consists on one visit).
  Interventions: Other: Immersive virtual reality task

INTERVENTIONS:
Other: Immersive virtual reality task — participants will have to wear a virtual reality headset connected to a remote control and will have to perform submersive virtual reality tasks

SUMMARY:
Spatial navigation is a high-level cognitive function allowing animals and humans to orient and move in space by constructing a mental representation of the environment. This function has been identified as one of the very first to be affected by Alzheimer's disease, including at the early stages, before the appearance of other mnesic disorders that the latter causes, such as those of episodic memory. However, the neuropsychological tests currently used in the diagnosis of cognitive disorders do not allow effective assessment of spatial memory impairment, in particular because it is impractical to offer spatial orientation tasks in a consulting room. In this context, virtual reality offers very interesting perspectives: it makes it possible to create controlled environments to assess spatial memory, without leaving the place of consultation.

Before being able to test its possible diagnostic efficacy, it is imperative to test the feasibility as well as the reliability of this type of task on an elderly population with no cognitive impairment. The data currently available on immersion tolerance in virtual reality mainly concern young people aged 18 to 35 and little data is available concerning the elderly or very old.

If this task correctly assesses spatial navigation abilities, this study should find the effects of age and sex usually observed.

The aim of this study is to assess the tolerance of an immersive virtual reality task evaluating the spatial memory of elderly subjects and the effects of age, gender and level of education on performance.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 60 to 85
* Participant affiliated or entitled to a social security scheme
* Recruited participants must have been informed and consented in writing

Exclusion Criteria:

* Participant with a diagnosis of cognitive impairment
* Severe, progressive or unstable pathology whose nature may interfere with the evaluation variables (epilepsy, psychiatric or psychotic disorders in the acute phase, visual hallucinations, acute infection, lack of sleep)
* Participant equipped with a pacemaker
* Burns or sores on the upper part of the face or on the scalp
* Consumption of toxic substances that can influence cognitive performance
* Deafness or blindness that may compromise participant assessment or completion of tasks and scales
* Participant under guardianship or curatorship or legal safeguard
* Participant refusing to use an immersive virtual reality tool
* Criterion for stopping the procedure under study: stopping the virtual reality task due to the participant's simulator sickness.
* Montreal Cognitive Assessment (MOCA) score less than 26
* MacNair Subjective Complaint Scale score greater than 16
* AGGIR score (Autonomy, Gerontology Group Iso Resources) less than 5

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Sickness Simulator Questionnaire (SSQ) score | The sickness simulator scale is assessed immediately after the immersive virtual reality task.
  This is a questionnaire composed of 16 items covering the potential symptoms of intolerance to a virtual reality tool.
  Each item is rated 0 (no symptom), 1 (mild symptom), 2 (moderate symptom) or 3 (severe symptom). The total score is obtained by multiplying the sum of the items by 3.74, and therefore varies from 0 to 180.

SECONDARY OUTCOMES:
Time to complete the task in immersive virtual reality according to the age of the participants | through study completion, 1 year
  Time to complete the task in immersive virtual reality (in seconds) according to the age of participants (in years)
Time to complete the task in immersive virtual reality (in seconds) according to the gender of participants (male or female) | through study completion, 1 year
  Time to complete the task in immersive virtual reality according to the gender of participants
Time to complete the task in immersive virtual reality according to the number of years of study | through study completion, 1 year
  Time to complete the task in immersive virtual reality (in seconds) according to the number of years of study (from entry into primary school)
Raw score on the Wechsler Memory Scale-III (MEM III) Spatial Memory subtest | through study completion, 1 year
  The test is designed for adults and the elderly to assess the performance of auditory memory, visual memory, memory immediate, delayed and visual working memory.The subtest used is the Spatial Memory subtest, it ranges from 0 to 28 (the higher the score, the better the performance).

CONTACTS AND LOCATIONS:
Locations (1):
- Charpennes Geriatric Hospital, Lyon University Hospital, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No